CLINICAL TRIAL: NCT03324945
Title: Chemotherapy-Induced Cognitive Impairment in Patients With Ovarian Cancer: A Phase II Study of the Cognitive Effects of Platinum/Taxane-based Chemotherapy in Patients With Ovarian Cancer
Brief Title: Chemotherapy-Induced Cognitive Impairment in Ovarian Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rachel Miller (Other)
Collaborators: Office of US Army Medical Research and Material Command (Unknown)
Responsible Party: Sponsor-Investigator, Rachel Miller, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-15-GYN-333
Record Dates: First submitted 2017-09-15; First posted 2017-10-30 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Chemotherapy-induced Cognitive Impairment
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurocognitive Assessment +/- FMRI (Experimental): All participants receive pre- and post-chemotherapy neurocognitive assessments. A sequentially-assigned subset also receive pre- and post-chemotherapy Functional Magnetic Resonance Imaging (FMRI) procedures.
  Interventions: Behavioral: Neurocognitive assessments

INTERVENTIONS:
Behavioral: Neurocognitive assessments — Baseline and post-chemotherapy neurocognitive testing. A sequentially-assigned subset of participants also receive baseline and post-chemotherapy neuroimaging (FMRI)

SUMMARY:
Chemotherapy-induced cognitive impairment (CICI), also known as "chemobrain," is a spectrum of neurocognitive deficits experienced during and after the administration of chemotherapy for cancer. The incidence of CICI is significant, affecting anywhere from 25 to 75% of survivors, and the biologic basis is unknown. This novel study is designed to address the questions of incidence and biological cause for CICI, while gaining a better understanding of the structural and functional effects of chemotherapy on the brain.

DETAILED DESCRIPTION:
Chemotherapy-induced cognitive impairment (CICI), also known as "chemobrain," is a spectrum of neurocognitive deficits experienced during and after the administration of chemotherapy for cancer. The incidence of CICI is significant, affecting anywhere from 25 to 75% of survivors, and the biologic basis is unknown. This novel study is designed to address the questions of incidence and biological cause for CICI, while gaining a better understanding of the structural and functional effects of chemotherapy on the brain. In order to address these important objectives, a diverse team of experienced investigators has been assembled to design and implement the proposed protocol. The research team for this project seeks to accomplish the proposed objectives through following mechanisms: 1) assessment of the neurocognitive domains affected in CICI using a tailored battery of cognitive tests to define CICI; 2) measurement of serum markers of oxidative stress and correlation of these markers with neurocognitive test results; and 3) exploration of structural and functional changes in the brain during cognitive tasks and correlation of results with markers of oxidative stress and neurocognitive test results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any stage epithelial ovarian cancer, including cancers arising from the fallopian tube and primary peritoneal cancer, or patients with other gynecologic malignancy (any stage), who are chemotherapy-naïve, and scheduled to undergo at least 6 cycles of intravenous platinum/taxane-based chemotherapy.
2. Patients must have adequate bone marrow, renal, hepatic, and sensory neurologic function to be eligible to receive platinum/taxane-based chemotherapy.
3. Patients must have a World Health Organization Performance Status of ≤ 2.
4. Age ≥18 years.
5. Ability to understand and the willingness to sign an approved written informed consent document.

Exclusion Criteria:

1. Patients who have received prior cytotoxic chemotherapy are ineligible. Patients may have received prior adjuvant hormonal therapy for localized breast cancer, provided that it was completed prior to registration, and that the patient remains free of recurrent or metastatic disease.
2. Patients undergoing neoadjuvant chemotherapy with planned interval cytoreductive surgery and adjuvant therapy are not included in this group.
3. Patients who are receiving any other investigational agents are excluded.
4. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic outcomes and other adverse events.
5. With the exception of non-melanoma skin cancer and other specific malignancies noted above, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last five years or whose previous cancer treatment contraindicates this therapy are excluded.
6. Patients with underlying dementia (or on medications to treat Alzheimer's disease such as donepezil, rivastigmine, galantamine, tacrine, or memantine), encephalopathy, or other neurological disorder known to adversely affect cognition (such as epilepsy or prior stroke) are excluded. (Patients with depression or anxiety are not excluded).
7. Patients will be excluded from fMRI testing if they are left-handed, claustrophobic, have a pacemaker, or have metal implants. Patients not undergoing fMRI testing may still enroll in clinical trial, including the ERP testing, if all other eligibility criteria are met.
8. Patients who are pregnant or nursing are excluded. Pregnant women are excluded from this study because cytotoxic chemotherapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cytotoxic chemotherapy, breastfeeding should be discontinued if the mother is treated with cytotoxic chemotherapy.
9. Patients who are non-English speaking are excluded because of the inability to adequately administer neurocognitive testing in non-English languages.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Reliable Change Index (RCI) | 4 weeks after completing cycle #6 chemotherapy (each cycle is 21 days)
  To address the primary aim, RCI (which is essentially a z-score) for each patient will be calculated from the pre-, post-chemotherapy Montreal Cognitive Assessment (MoCA) test results. Then a Wilcoxon signed rank test will be applied to the RCI values with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Assess the correlation between biologic markers of oxidative stress and neurocognitive test results. | 4 weeks after completing cycle #6 chemotherapy (each cycle is 21 days)
  Analysis of covariance (ANCOVA), adjusting for baseline log serum levels, will be utilized to assess for differences in log levels over timepoints including the 4 and 6 hour samples. Spearman correlations will be utilized to describe associations with cognitive tests scores and biochemical measured in addition to Spearman Correlation coefficients between baseline biochemical measures.
Assess the correlation between brain imaging and neurocognitive test results | 4 weeks after completing cycle #6 chemotherapy (each cycle is 21 days)
  For neurological outcomes, a longitudinal comparison before and after Chemotherapy in fMRI (percent signal change and extend of activation voxels), DTI (FA % change), and ERP (uV) will be performed. There will be changes in patterns of fMRI responses, FA, and ERP signals from baseline to after treatment. We expect that fMRI activation will be change in prefrontal regions change of effort needed to do the memory task. Changes in white matter FA in after the treatment may be observable in the white matter regions such as the frontal and temporal cortices as well as in gray matter regions suspected to be affected by the Chemo. Cognitive ERP patterns will be changed in the same individuals. fMRI and ERP analysis can be analyzed and compared at individual level.
  To explore correlations between fMRI outcomes and cognitive measures, ANCOVA is an appropriate choice since we want to study measures after treatment, relative to initial values.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel W Miller, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No